CLINICAL TRIAL: NCT01816425
Title: Comparison Between Cobalt-chromium Partial Dentures and Thermoplastic Partial Dentures: Random Clinical Trial
Brief Title: Comparison Between Cobalt-chromium Partial Dentures and Thermoplastic Partial Dentures
Acronym: Flex
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Érico Castaldin Fraga Moreira, Master of Science, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Thermoplastic Denture Base
Record Dates: First submitted 2013-02-20; First posted 2013-03-22 (Estimated); Last update posted 2013-03-25 (Estimated); Status verified 2013-03

CONDITIONS: Jaw, Edentulous, Partially
Keywords: Dental Prosthesis; Dental Prosthesis Design
MeSH Terms: conditions — Jaw, Edentulous, Partially

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- thermoplastic partial denture (Experimental): The patients that need oral rehabilitation with partial denture will receive a thermoplastic partial denture as treatment
  Interventions: Device: Thermoplastic partial denture
- CoCr partial denture (Active Comparator): The patients that need oral rehabilitation with partial denture will receive a CoCr partial denture as treatment
  Interventions: Device: CoCr partial denture

INTERVENTIONS:
Device: Thermoplastic partial denture
  Arms: thermoplastic partial denture
Device: CoCr partial denture
  Arms: CoCr partial denture

SUMMARY:
The cobalt-chromium (CoCr) partial denture has been made for a long period. It respects biomechanical principles, providing harmony between mechanical and biological activities. The fundamental principles of biomechanics applied in the manufacture of steel structure are: retention, reciprocity, attachment and stability. To get the proper planning, we need to assess the dental support system, with its qualitative and quantitative values. But conventional dentures has a inherent problem which is the metallic elements apparent and in some cases the stiffness of the component support elements that generates stress.

The Thermoplastic partial dentures increase aesthetics in replacement of metal structures in oral rehabilitation. So many treatments are being done in everyday practice without a defined concept on various aspects of its construction and oral applicability.

This trial aims to assess the basic parameters of both dentures in: nutrition, speech therapy, chewing force, chewing efficiency and quality of life.

60 years old or older patients who require removable prosthesis. These will be randomly selected for the fabrication and installation of removable partial dentures (Gold Standard - control group - CoCr partial denture) and thermoplastic partial denture(experimental group).

Before beginning the work, selected patients will make some preliminary tests such as controlling the individual condition, they are:

* three questionnaires:
* instrument for assessing quality of life related to oral health, GOHAI - General Oral Health Assessment Index of Atchinson & Dolan
* instrument for assessing the social and economic profile of ABEP (Brazilian Association of Research Companies) CCEB 2011;
* Instrument for assessing cognitive condition MINI-MENTAL;
* Speech evaluation
* Nutritional assessment;
* Evaluation of masticatory efficiency and
* Chewing strength. After preliminary assessments patients will be subjected to treatments for manufacture of partial dentures. After the installation (end of the technical construction of the dentures) and the adjustments appointment the tests will be repeated and in successive control periods of 3 months, 6 months, 12 months, 18 months and 24 months respectively, when the tests will do again now to see if there was a change in the initial condition.

ELIGIBILITY:
Inclusion Criteria:

60 years old or older patient with partial edentulous jaws with indication of removable partial denture

Exclusion Criteria:

patient younger than 60 years patient with edentulous mouth

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-02; Primary Completion 2013-11 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Comparison between thermoplastic partial denture and CoCr partial dentures | 24 months
  the tests result of the thermoplastic partial denture will be compared with the tests result of the CoCr partial dentures, the hypothesis is that thermoplastic partial denture are similar to CoCr partial dentures

CONTACTS AND LOCATIONS:
Overall Officials: Roberto C Stegun, Phd, Principal Investigator — Dentistry College, University of São Paulo
Locations (1):
- Dentistry College, University of São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] VandenBrink JP, Wolfaardt JF, Faulkner MG. A comparison of various removable partial denture clasp materials and fabrication procedure for placing clasps on canine and premolar teeth. J Prosthet Dent. 1993 Aug;70(2):180-8. doi: 10.1016/0022-3913(93)90016-h. PMID 8103801
- [Background] Wu JC, Latta GH Jr, Wicks RA, Swords RL, Scarbecz M. In vitro deformation of acetyl resin and metal alloy removable partial denture direct retainers. J Prosthet Dent. 2003 Dec;90(6):586-90. doi: 10.1016/j.prosdent.2003.09.020. PMID 14668760